CLINICAL TRIAL: NCT01147822
Title: A Study to Evaluate Efficacy and Safety of Pazopanib Versus Sunitinib for the Treatment of Asian Subjects With Locally Advanced and/or Metastatic Renal Cell Carcinoma - A Substudy to VEG108844
Brief Title: Pazopanib Versus Sunitinib in the Treatment of Asian Subjects With Locally Advanced and/or Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113078; CPZP034A2201 (Other: Novartis); VEG113078 (Other: GlaxoSmithKline)
Record Dates: First submitted 2010-05-20; First posted 2010-06-22 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: SUTENT; GW76034; Sunitinib; Renal cell carcinoma; Pazopanib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pazopanib (Experimental): 800 mg administered once daily orally continuous dosing
  Interventions: Drug: Pazopanib
- Sunitinib (Active Comparator): 50 mg sunitinib to be administered in 6-week cycles: 50 mg orally daily for 4 weeks followed by 2 weeks off treatment
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Pazopanib — 800 mg administered once daily orally continuous dosing
  Other Names: GW786034
  Arms: Pazopanib
Drug: Sunitinib — 50 mg sunitinib to be administered in 6-week cycle: 50 mg orally daily for 4 weeks followed by 2 weeks off treatment
  Arms: Sunitinib

SUMMARY:
This was a randomized, open label, parallel group, Phase II study to evaluate the efficacy and safety of pazopanib compared to sunitinib in Asian subjects with advanced renal cell carcinoma (RCC) who have not received prior systemic therapy for advanced or metastatic RCC.

DETAILED DESCRIPTION:
Study VEG113078 is a substudy of Study VEG108844 (NCT00720941). Due to the projected limited enrollment of Asian participants into Study VEG108844, Study VEG113078 was designed to evaluate the efficacy and safety of pazopanib versus sunitinib for the treatment of Asian participants enrolled from selected Far-East Asian countries. The data for Study VEG113078 was pooled at the same time as the main study VEG108844 (NCT00720941). The subjects were centrally randomized in 1:1 ratio to receive open label study medication of either pazopanib 800mg to be administered once daily orally continuous dosing or sunitinib 50mg to be administered in 6-week cycles: 50mg orally daily for 4 weeks followed by 2 weeks off treatment. Subjects were permitted to receive supportive care throughout the study including transfusion of blood and blood products, treatment with antibiotics, anti-emetics, anti-diarrheal agents, analgesics, erythropoietin, or bisphosphonates, when appropriate. The study treatment continued until subjects experience disease progression, unacceptable toxicity, withdraw consent, or death.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of renal cell carcinoma with clear-cell component histology.
* Received no prior systemic therapy (interleukin-2, interferon-alpha, chemotherapy, bevacizumab, mTOR inhibitor, sunitinib, sorafenib or other VEGF TKI) for advanced or metastatic RCC
* Locally advanced or metastatic renal cell carcinoma Measurable disease by CT or MRI
* Karnofsky performance scale status of >=70
* Age >=18 years
* A female is eligible to enter and participate in this study if she is of: non-childbearing or agrees to use adequate contraception.
* Adequate organ system function
* Total serum calcium concentration <12.0mg/dL
* Left ventricular ejection fraction >= lower limit of institutional normal

Exclusion Criteria:

* Pregnant or lactating female (unless agrees to refrain from nursing throughout the treatment period and for 14 days following the last dose of study)-History of another malignancy (unless have been disease-free for 3 years)
* History or clinical evidence of central nervous system (CNS) metastases (unless have previously-treated CNS metastases and meet all 3 of the following criteria are: are asymptomatic, have had no evidence of active CNS metastases for >=6 months prior to enrolment, and have no requirement for steroids or enzyme-inducing anticonvulsants)
* Clinically significant gastrointestinal abnormalities including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug, active peptic ulcer disease, known intraluminal metastatic lesion/s with suspected bleeding, Inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Presence of uncontrolled infection
* Prolongation of corrected QT interval (QTc) > 480 milliseconds
* History of any one or more of the following cardiovascular conditions within the past 12 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association
* History of cerebrovascular accident including transient ischemic attack within the past 12 months
* History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months (unless had recent DVT and have been treated with therapeutic anti-coagulating agents for at least 6 weeks)
* Poorly controlled hypertension (defined as systolic blood pressure of >=150mmHg or diastolic blood pressure of >=90mmHg). Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding susceptibility
* Spitting/coughing up blood within 6 weeks of first dose of study drug
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study
* Use any prohibited medications within 14 days of the first dose of study medication
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug
* Prior use of an investigational or licensed drug that targets VEGF or VEGF receptors (eg. bevacizumab, sunitinib, sorafenib, etc), or are mTOR inhibitors (eg. temsirolimus, everolimus, etc).
* Is now undergoing and/or has undergone in the 14 days immediately prior to first dose of study drug, any cancer therapy (surgery, tumor embolization, chemotherapy, radiation therapy, immunotherapy, biological therapy, or hormonal therapy)
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or sunitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- China (6):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- South Korea (3):
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Goyang-si, Gyeonggi-Do
  - Novartis Investigative Site, Seoul
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung Hsien
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sheng X, Jin J, He Z, Huang Y, Zhou A, Wang J, Ren X, Ye D, Zhang X, Qin S, Zhou F, Wang B, Guo J. Pazopanib versus sunitinib in Chinese patients with locally advanced or metastatic renal cell carcinoma: pooled subgroup analysis from the randomized, COMPARZ studies. BMC Cancer. 2020 Mar 14;20(1):219. doi: 10.1186/s12885-020-6708-8. PMID 32171288
- [Derived] Guo J, Jin J, Oya M, Uemura H, Takahashi S, Tatsugami K, Rha SY, Lee JL, Chung J, Lim HY, Wu HC, Chang YH, Azad A, Davis ID, Carrasco-Alfonso MJ, Nanua B, Han J, Ahmad Q, Motzer R. Safety of pazopanib and sunitinib in treatment-naive patients with metastatic renal cell carcinoma: Asian versus non-Asian subgroup analysis of the COMPARZ trial. J Hematol Oncol. 2018 May 22;11(1):69. doi: 10.1186/s13045-018-0617-1. PMID 29788981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 58 centers in 4 countries in Asia (China, Korea, Taiwan, and Japan).
Pre-assignment Details: Participants were stratified based on Karnofsky Performance Scale scores (70 or 80; 90 or 100), Baseline levels of lactate dehydrogenase (>1.5 versus <=1.5 times the upper limit of normal [ULN]), and previous nephrectomy (yes versus no) and were randomized in a 1:1 ratio to receive either pazopanib or sunitinib.
Groups:
- Pazopanib 800 mg: Participants were administered pazopanib 800 milligrams (mg) (2 x 400 mg tablets) orally once daily (OD) continuously. Pazopanib was to be taken at least one hour before or at least two hours after a meal. Study treatment continued until participants experienced disease progression, death, or unacceptable toxicity, or withdrew consent for any other reason.
- Sunitinib 50 mg: Participants were administered sunitinib 50 mg capsules orally OD in 6-week cycles (4 weeks of treatment, followed by 2 weeks without treatment). Study treatment continued until participants experienced disease progression, death, or unacceptable toxicity, or withdrew consent for any other reason.
Period: Overall Study
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Started (All Asian randomized subjects were included in the Intent-to-Treat (ITT) Population) | 188 | 179
Safety Population (All Asian randomized subjects who received at least one dose of study treatment were included in the Safety Population) | 186 | 177
Completed | 150 | 143
Not Completed | 38 | 36
Not completed — Lost to Follow-up | 14 | 6
Not completed — Withdrawal by Subject | 10 | 16
Not completed — Physician Decision | 9 | 8
Not completed — Transitioned to another mechanism of continuing pazopanib or sunitinib therapy after 30SEP2013 | 4 | 5
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg | Total
Number analyzed (Participants) | 188 | 179 | 367
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (11.51) | 57.6 (11.19) | 57.6 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 42 | 93
  Male | 137 | 137 | 274
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Central/South Asian Heritage | 2 | 1 | 3
  Asian - East Asian Heritage | 154 | 144 | 298
  Asian - Japanese Heritage | 29 | 31 | 60
  Asian - South East Asian Heritage | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval between the date of randomization and the earliest date of progressive disease (PD), as defined by the Independent Review Committee (IRC), or death due to any cause. The IRC defined PD per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1. Per RECIST, PD is defined as a >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of >=1 new lesion.
Time Frame: From randomization until the earliest date of disease progression or date of death from any cause, assessed up to approximately 24 months (Primary analysis cut-off date = 21-May-2012) at the same time as the main study VEG108844 (NCT00720941).
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Participants who had neither progressed nor died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 188 | 179
Months | 8.4 [8.3 to 11.1] | 11.1 [8.2 to 14.3]
Statistical Analysis 1: Comparison: Pazopanib 800 mg vs Sunitinib 50 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 1.0184, 95% CI 2-sided [0.7658 to 1.3542] — The HR was estimated by the Cox regression model using treatment stratification factors as covariates. The HR was adjusted for Karnofsky Performance Scale scores, prior nephrectomy, and Baseline levels of lactate dehydrogenase

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time (in months) from the date of randomization to the date of death due to any cause. If the patient was not known to have died, then OS was censored. The censoring date was date of the last study visit, or contact, until the cut-off date. The cut-off date was not used for last contact date, unless the patient was seen or contacted on that date.
Time Frame: From randomization until date of death from any cause, assessed up to 40 months (Final OS analysis cut-off date = 30-Sep-2013) at the same time as the main study VEG108844 (NCT00720941).
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Participants who had not died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 188 | 179
Months | 26.7 [23.7 to 41.7] | 33.4 [26.9 to 39.6]
Statistical Analysis 1: Comparison: Pazopanib 800 mg vs Sunitinib 50 mg; Test type: Superiority or Other; p = 0.604, Log Rank; Hazard Ratio (HR) = 1.080, 95% CI 2-sided [0.808 to 1.441] — Hazard ratios were estimated using the Pike estimator. A hazard ratio <1 indicates a lower risk with this treatment compared with Sunitinib

3. Secondary Outcome: Overall Response Rate (ORR) as Assessed by Independent Review
Description: Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline per central review assessment.
Time Frame: From randomization until date of radiographic progression, assessed up to approximately 24 months (Primary analysis cut-off date = 21-May-2012) at the same time as the main study VEG108844 (NCT00720941).
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 188 | 179
Percentage of Participants | 36 [28.8 to 42.5] | 21 [14.7 to 26.6]

4. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the start of treatment until the first documented evidence of CR (the disappearance of all target and non-target lesions) or PR (at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD), whichever comes first. CR and PR were evaluated by an independent review per RECIST, Version 1.
Time Frame: as for outcome 3
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Only those participants who experienced either a confirmed CR or a PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 67 | 37
Weeks | 11.9 [6.7 to 12.3] | 17.9 [12.0 to 23.9]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented evidence of response (CR or PR) until the first documented sign of disease progression (a >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of >=1 new lesion) or death, if sooner. CR=the disappearance of all target and non-target lesions. PR=at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD.
Time Frame: From the date of the first documented response (CR or PR) to the date of first documented progression, assessed up to approximately 24 months (Primary analysis cut-off date = 21-May-2012) at the same time as the main study VEG108844 (NCT00720941).
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Only those participants who had either a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 67 | 37
Months | 15.2 [9.9 to 17.9] | 18.0 [12.3 to NA] — An insufficient number of responders were followed until progression to observe the end of response; thus, the upper limit of the confidence interval could not be calculated.

6. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from first dose of study medication to 28 days after last dose of study medication (on-treatment), up to approximately 125 months.
  Deaths were collected in the post treatment survival follow up from 29 days after last dose of study medication until the end of the study, up to approximately 135 months.
Time Frame: Pre-treatment deaths: Up to 21 days prior to treatment. On-treatment deaths: Up to 125 months. Post-treatment deaths: up to 135 months.
Population: Intent-to-Treat (ITT) Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 188 | 179
Participants
  Pre-treatment deaths | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 186 | 177
  On-treatment deaths | 7 | 6
  Post-treatment deaths: number analyzed (Participants) | 179 | 171
  Post-treatment deaths | 92 | 80
  All deaths | 99 | 86

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 28 days post-treat follow-up, assessed up to approximately 125 months. Deaths were recorded from study start date until end of survival follow-up phase (end of study), assessed up to approximately 135 months.
Description: Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Pazopanib 800 mg: Pazopanib 800 mg: Events up to 28 days post-treatment
- Sunitinib 50 mg: Sunitinib 50 mg: Events up to 28 days post-treatment
- Pazopanib 800 mg (Post-Treatment): Pazopanib 800 mg (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Sunitinib 50 mg (Post-Treatment): Sunitinib 50 mg (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg | Pazopanib 800 mg (Post-Treatment) | Sunitinib 50 mg (Post-Treatment)
All-Cause Mortality (participants affected / at risk) | 7/188 | 6/179 | 92/179 | 80/171
Serious Adverse Events (participants affected / at risk) | 76/186 | 76/177 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 182/186 | 173/177 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=186) | Sunitinib 50 mg (N=177) | Pazopanib 800 mg (Post-Treatment) (N=0) | Sunitinib 50 mg (Post-Treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 15 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | NA | NA
Angina unstable (Cardiac disorders) | 1 | 1 | NA | NA
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | NA | NA
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | NA | NA
Myocardial infarction (Cardiac disorders) | 1 | 1 | NA | NA
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | NA | NA
Anal fistula (Gastrointestinal disorders) | 1 | 0 | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 0 | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | NA | NA
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | NA | NA
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastritis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Ileus (Gastrointestinal disorders) | 2 | 0 | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | NA | NA
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 0 | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | NA | NA
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | NA | NA
Asthenia (General disorders) | 0 | 3 | NA | NA
Disease progression (General disorders) | 1 | 0 | NA | NA
Fatigue (General disorders) | 1 | 4 | NA | NA
Pain (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 3 | 6 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 3 | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | NA | NA
Appendicitis (Infections and infestations) | 1 | 1 | NA | NA
Cellulitis (Infections and infestations) | 1 | 0 | NA | NA
Complicated appendicitis (Infections and infestations) | 0 | 1 | NA | NA
Gastroenteritis (Infections and infestations) | 0 | 1 | NA | NA
H1N1 influenza (Infections and infestations) | 1 | 0 | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | NA | NA
Infection (Infections and infestations) | 1 | 0 | NA | NA
Perinephric abscess (Infections and infestations) | 0 | 1 | NA | NA
Peritonitis (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 4 | 1 | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 1 | NA | NA
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | NA | NA
Septic shock (Infections and infestations) | 1 | 0 | NA | NA
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Alanine aminotransferase increased (Investigations) | 11 | 3 | NA | NA
Amylase increased (Investigations) | 0 | 1 | NA | NA
Aspartate aminotransferase increased (Investigations) | 4 | 0 | NA | NA
Blood bilirubin increased (Investigations) | 1 | 1 | NA | NA
Blood calcium increased (Investigations) | 0 | 1 | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | NA | NA
Blood glucose decreased (Investigations) | 1 | 0 | NA | NA
Blood magnesium decreased (Investigations) | 0 | 1 | NA | NA
Blood potassium increased (Investigations) | 1 | 0 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | NA | NA
Lipase increased (Investigations) | 4 | 3 | NA | NA
Liver function test abnormal (Investigations) | 1 | 0 | NA | NA
Neutrophil count decreased (Investigations) | 2 | 0 | NA | NA
Platelet count decreased (Investigations) | 0 | 7 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1 | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | NA | NA
Cerebral infarction (Nervous system disorders) | 0 | 2 | NA | NA
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | NA | NA
Dizziness (Nervous system disorders) | 0 | 1 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | NA | NA
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | NA | NA
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | NA | NA
Syncope (Nervous system disorders) | 0 | 1 | NA | NA
Tremor (Nervous system disorders) | 0 | 1 | NA | NA
Mental status changes (Psychiatric disorders) | 1 | 0 | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 1 | NA | NA
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | NA | NA
Arterial rupture (Vascular disorders) | 0 | 1 | NA | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | NA | NA
Hypertension (Vascular disorders) | 1 | 1 | NA | NA
Hypertensive crisis (Vascular disorders) | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=186) | Sunitinib 50 mg (N=177) | Pazopanib 800 mg (Post-Treatment) (N=0) | Sunitinib 50 mg (Post-Treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 11 | 50 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 40 | 61 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 3 | 11 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 43 | 77 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 29 | 80 | NA | NA
Hyperthyroidism (Endocrine disorders) | 3 | 11 | NA | NA
Hypothyroidism (Endocrine disorders) | 31 | 55 | NA | NA
Eyelid oedema (Eye disorders) | 17 | 29 | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 12 | 17 | NA | NA
Abdominal distension (Gastrointestinal disorders) | 11 | 14 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 18 | 18 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 29 | 23 | NA | NA
Constipation (Gastrointestinal disorders) | 14 | 33 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 103 | 81 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 19 | 24 | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 6 | 10 | NA | NA
Mouth ulceration (Gastrointestinal disorders) | 17 | 26 | NA | NA
Nausea (Gastrointestinal disorders) | 44 | 42 | NA | NA
Stomatitis (Gastrointestinal disorders) | 25 | 55 | NA | NA
Toothache (Gastrointestinal disorders) | 5 | 11 | NA | NA
Vomiting (Gastrointestinal disorders) | 41 | 29 | NA | NA
Asthenia (General disorders) | 8 | 9 | NA | NA
Face oedema (General disorders) | 10 | 33 | NA | NA
Fatigue (General disorders) | 82 | 91 | NA | NA
Mucosal inflammation (General disorders) | 12 | 20 | NA | NA
Oedema (General disorders) | 8 | 20 | NA | NA
Oedema peripheral (General disorders) | 13 | 20 | NA | NA
Pyrexia (General disorders) | 20 | 25 | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 17 | 10 | NA | NA
Gingivitis (Infections and infestations) | 12 | 8 | NA | NA
Nasopharyngitis (Infections and infestations) | 16 | 19 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 11 | 12 | NA | NA
Alanine aminotransferase increased (Investigations) | 71 | 55 | NA | NA
Amylase increased (Investigations) | 25 | 16 | NA | NA
Aspartate aminotransferase increased (Investigations) | 71 | 58 | NA | NA
Bilirubin conjugated increased (Investigations) | 17 | 6 | NA | NA
Blood albumin decreased (Investigations) | 12 | 15 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 19 | 12 | NA | NA
Blood bilirubin increased (Investigations) | 34 | 26 | NA | NA
Blood bilirubin unconjugated increased (Investigations) | 16 | 8 | NA | NA
Blood cholesterol increased (Investigations) | 12 | 16 | NA | NA
Blood creatinine increased (Investigations) | 32 | 52 | NA | NA
Blood glucose increased (Investigations) | 10 | 13 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 27 | 45 | NA | NA
Blood phosphorus decreased (Investigations) | 9 | 11 | NA | NA
Blood thyroid stimulating hormone increased (Investigations) | 18 | 31 | NA | NA
Blood triglycerides increased (Investigations) | 18 | 24 | NA | NA
Blood urea increased (Investigations) | 10 | 14 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 18 | 7 | NA | NA
Haematocrit decreased (Investigations) | 6 | 12 | NA | NA
Haemoglobin decreased (Investigations) | 22 | 50 | NA | NA
Lipase increased (Investigations) | 22 | 19 | NA | NA
Neutrophil count decreased (Investigations) | 22 | 46 | NA | NA
Platelet count decreased (Investigations) | 30 | 58 | NA | NA
Protein total decreased (Investigations) | 8 | 9 | NA | NA
Red blood cell count decreased (Investigations) | 2 | 10 | NA | NA
Weight decreased (Investigations) | 19 | 5 | NA | NA
White blood cell count decreased (Investigations) | 27 | 54 | NA | NA
Xanthochromia (Investigations) | 1 | 11 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 78 | 69 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 15 | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 9 | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 11 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 11 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 8 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 17 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 18 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 16 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 20 | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 10 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 13 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 19 | NA | NA
Dizziness (Nervous system disorders) | 18 | 18 | NA | NA
Dysgeusia (Nervous system disorders) | 11 | 15 | NA | NA
Headache (Nervous system disorders) | 27 | 23 | NA | NA
Hypogeusia (Nervous system disorders) | 9 | 13 | NA | NA
Taste disorder (Nervous system disorders) | 14 | 23 | NA | NA
Insomnia (Psychiatric disorders) | 10 | 15 | NA | NA
Haematuria (Renal and urinary disorders) | 8 | 12 | NA | NA
Proteinuria (Renal and urinary disorders) | 61 | 54 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 26 | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 20 | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 29 | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 11 | NA | NA
Hair colour changes (Skin and subcutaneous tissue disorders) | 67 | 15 | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 93 | 114 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 16 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 27 | 37 | NA | NA
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 15 | 5 | NA | NA
Yellow skin (Skin and subcutaneous tissue disorders) | 4 | 42 | NA | NA
Hypertension (Vascular disorders) | 103 | 94 | NA | NA

LIMITATIONS AND CAVEATS:
This is a legacy GlaxoSmithKline (GSK) study and the primary CSR was completed by GSK prior to the study sponsorship handover. The full investigators lists and other appendices were not transferred over during the change in sponsorship from GSK to Novartis and therefore, the team could not confirm or quality control the investigator sites list.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.